CLINICAL TRIAL: NCT05701722
Title: Effects of Flourish HEC Vaginal Care System on Vaginal Microbiome in Women With Recurrent Bacterial Vaginosis
Brief Title: Effect of Flourish HEC Vaginal Care System on BV Recurrence and the Vaginal Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vaginal Biome Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BV30123
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Bacterial Vaginosis
Keywords: vaginal microbiome; vaginal pH; Probiotic; Lactobacillus
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine Care (No Intervention): Women with recurrent BV who are randomly assigned to the Routine Care (control) arm will undergo assessments at baseline, 12 weeks, and 24 weeks. They will be treated with appropriate antibiotics or antifungals in case of BV or yeast infection, respectively, but otherwise will not receive any treatment. They may engage in any vulvovaginal hygiene of their choosing except for using products made by Good Clean Love.
- Flourish HEC (Experimental): Women with recurrent BV who are randomly assigned to the Flourish HEC (intervention) arm will undergo assessments at baseline, 12 weeks, and 24 weeks. They will receive routine care as needed (see Routine Care arm). In addition, they will use the Flourish HEC Vaginal Care System regularly for the 24-week duration of the study. Briefly, they will use Balance intimate wash daily with regular bathing; BioNourish vaginal moisturizing gel every other day; and BiopHresh homeopathic vaginal suppository with probiotics every 3rd day. They will use no other products (except menstrual hygiene products) in the vulvovaginal area during the study.
  Interventions: Device: Flourish HEC Vaginal Care System

INTERVENTIONS:
Device: Flourish HEC Vaginal Care System — BioNourish, a component of the Flourish HEC system, is a class II medical device. In addition to BioNourish, the system includes Balance intimate wash and BiopHresh homeopathic vaginal suppository with probiotics. All products are available over the counter and have been on the market for several years.
  Other Names: BioNourish Vaginal Moisturizing Gel
  Arms: Flourish HEC

SUMMARY:
The goal of this clinical trial is to learn about the vaginal microbiome in premenopausal women with recurrent bacterial vaginosis (BV). The main questions it aims to answer are:

* Does using a specific vaginal care system reduce recurrence of BV?
* How does using this vaginal care system change the vaginal microbiome and pH over time?

Participants will:

* Have their vaginal microbiome and pH tested in several ways at three timepoints: the start of the study, 12 weeks later, and 24 weeks after the start of the study
* Answer questionnaires about vulvovaginal symptoms at each of these three timepoints
* Use a specific vaginal care system at home for 24 weeks, consisting of an intimate wash, a vaginal moisturizing gel, and a vaginal probiotic suppository, if assigned to the intervention group

Researchers will compare the group using the vaginal care system with a control group that does not use the system to see if using the system reduces risk of BV recurrence or changes the vaginal microbiome, pH, or symptoms.

DETAILED DESCRIPTION:
The vaginal microbiome interacts with vaginal epithelial cells and host immune cells in varying ways depending on the presence of particular species. Presence of high quantities of Lactobacillus species, which are considered healthy, downregulate pro-inflammatory markers and upregulate anti-inflammatory markers. On the other hand, BV-associated bacteria such as Gardnerella vaginalis, Atopobium (Fannyhessea) vaginae, Prevotella bivia, Mobiluncus curtisii and others, are associated with increased pro-inflammatory markers and reduced anti-inflammatory molecules. The investigators predict that improving the vaginal microbiome by using an over-the-counter vaginal care system will increase levels of Lactobacillus species, reduce levels of BV-associated bacteria, and improve vulvovaginal symptoms of BV.

Bacterial vaginosis (BV) is a common dysbiosis of the vaginal microbiome causing vaginal odor, discharge, discomfort, or even vulvovaginal pain. In some women, BV is asymptomatic; there is some evidence to support the concept that asymptomatic BV results from repeated instances of BV that damage the vaginal lining so extensively that the body is no longer able to generate symptoms, and as such, asymptomatic BV represents a more advanced disease state as compared with symptomatic BV. Whether symptomatic or asymptomatic, BV is known to affect the vaginal epithelium, disrupting intercellular adhesions and increasing susceptibility to infections, including HIV, HSV, and perinatal infections leading to sequelae such as late miscarriage, preterm labor, preterm premature rupture of membranes, and preterm delivery. Symptomatic BV can interfere profoundly with quality of life, causing embarrassment, itching, pain, and challenges with intimacy. The standard of care for treatment of BV is metronidazole, clindamycin, or rarely other antibiotic. Repeated use of antibiotics is used out of necessity for symptomatic women, but many women and healthcare providers are hesitant to use antibiotics repeatedly due to side effects and risk of development of antibiotic-resistant organisms. An alternative method of preventing and/or treating BV is therefore desirable.

An 11-week pilot study of similar, though less informative, design was recently conducted. Women with recurrent BV were recruited to use the Flourish® Vaginal Care System [using aloe-based Restore gel instead of hydroxyethylcellulose (HEC)-based BioNourish gel which is part of the Flourish HEC Vaginal Care System] for 11 weeks. Primary outcomes were vaginal fluid pH and whether or not women had BV recurrence. By the end of the study, the average vaginal fluid pH had fallen from mean (SD) of 4.54 (0.53) at week 0 to 4.08 (0.40) at week 11. At baseline, 30% of women had active BV. (These women were treated with standard of care oral metronidazole). The number of BV-positive women steadily declined until 5 weeks, at which point no woman had BV. There was no recurrence of BV in any woman through the end of the study.

Although this 11-week study is promising, the short time frame provides only limited information about BV recurrence, and there was no control group included. However, considering what has been published, we might have expected up to half of the women to have had a recurrence of BV during this time. By developing this new randomized controlled study with a longer time frame, we will have more certainty about whether prevention of BV recurrence is a feasible aim for a double-blind placebo-controlled randomized controlled trial in the future.

The present study will also expand upon the previous trial by providing data about the vaginal microbiome of women before and after use of the Flourish HEC Vaginal Care System. Historically, Amsel criteria (presence of 3 out of 4 of: thin grayish-white discharge, positive whiff test with addition of KOH to vaginal fluid, vaginal pH >4.5, and presence of >20% clue cells on wet mount microscopy of vaginal smear) or Nugent scoring (scoring method based on Gram stained vaginal fluid) were used to diagnose BV. More recently, existing data about changes in the vaginal microbiome during BV have been used to develop the commonly used clinical BV tests such as Aptima BV test (Hologic), SureSwab BV and Vaginitis test (Quest Diagnostics), Affirm VPIII test (BD Diagnostics), and others. Recently, next-generation sequencing (NGS) has been used to examine more thoroughly the complement of bacteria found in women with or without symptomatic BV. These studies shed some light on what would constitute a healthy microbiome if the Flourish HEC Vaginal Care System is successful at establishing a healthy colony of lactobacilli. However, the investigators are not aware of any studies that have examined changes in the entire vaginal microbiome using NGS before and after use of a vaginal probiotic suppository. This is important because the pre-NGS techniques used are limited in their ability to detect species. Some bacteria are resistant to traditional culture techniques and may have been missed in earlier culture-based studies. PCR-based tests are limited because they are used to assess presence or amount of specific targets which have been selected using information from culture-based studies. The Evvy Vaginal Microbiome Test using metagenomic sequencing, a type of NGS technology, is superior because it is able to detect every bacterial and fungal species present at a level of 0.1% of the microbiome or higher. Only rare species would be missed. While these rare species may be important for seeding following events that disrupt the vaginal microbiome (like antibiotic use), they likely have a small effect on day-to-day health.

A 2019 meta-analysis found that vaginal probiotics for BV are safe and effective, though the authors noted a need for studies with larger numbers of women. Similarly, a Cochrane review noted there is insufficient evidence for or against recommending use of vaginal probiotic in BV, and recommended larger, well-designed trials. One study that pre-dates next-generation sequencing found that use of a Lactobacillus acidophilus probiotic vaginal suppository was effective at treating BV but only until a woman's next menses. A randomized, placebo-controlled trial providing two species of Lactobacillus for two months showed that the probiotic restored a normal microbiome in women who used the supplement, but not in controls. It did not follow women beyond the end of the study, but interestingly, the authors suggested that an at-home kit - similar to the one used in the present study - would allow women to take control of their own health. The present study has a six-month time period and has the additional advantage over all other studies that the probiotic is part of a larger system that restores vaginal pH to the correct level to allow for growth of Lactobacillus spp., and to suppress growth of pathogens. This pH adjustment is accomplished with the use of racemic lactic acid, which has been shown to be important for vaginal health vs. use of only L-lactic acid. We believe this is the first randomized controlled study of a vaginal probiotic suppository which also encourages growth of those bacteria by establishing a healthy vaginal luminal environment.

The original Flourish® Vaginal Care System, with slightly different vaginal moisturizer (with aloe), has recently been shown in a clinical study to reduce vaginal pH from 4.81 (unhealthy, elevated) to 4.05 (healthy) and prevent recurrence of bacterial vaginosis over a 10-week study period1. The proposed study uses a newly formulated product that is gentler (no aloe) because the study population is likely to have high sensitivity based on inclusion criteria involving tissue trauma.

The investigators hypothesize that regular use of the Flourish HEC Vaginal Care System can improve the vaginal microbiome and lower vaginal pH, which will thereby prevent recurrence of bacterial vaginosis in women with recurrent BV and improve their vulvovaginal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Cis-gender women between ages 18 and 52
2. Premenopausal
3. Clinically diagnosed with BV twice in the past six months or three times within the past year (by provider-determined criteria)

Exclusion Criteria:

1. Known allergies or sensitivities to any ingredients of the Flourish HEC Vaginal Care System
2. Immunosuppressed or otherwise immunocompromised
3. Vaginal infection at the start of the study other than bacterial vaginosis or yeast infection (these may be treated prior to starting the protocol)
4. Recent (within past 3 months) use of any antibiotics except for treating BV
5. Surgery within the past 3 months
6. Pregnant or trying to conceive during the trial
7. Lactating women
8. Recent (within past 3 months) usage of any Good Clean Love® (GCL) products
9. Sexual trauma history causing psychiatric or mental health disorders which may be triggered by questions related to vulvar or vaginal health, by pelvic exams, or self-application of vaginal products

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Recurrence of bacterial vaginosis (BV) | 24 week duration of the study
  The number of separate BV episodes will be assessed between baseline and 24 weeks in each arm separately. BV may be diagnosed by clinical test (Aptima, SureSwab, Affirm VPIII, etc.) that is routinely used by the study site; Amsel criteria; and/or Nugent scores. Where there is discordance between tests, the participant will be BV positive if 2/3 tests are positive. BV positive by Amsel criteria include having at least 3 of the following 4 parameters: 1) thin, white-to-gray homogeneous vaginal discharge; 2) amine odor upon addition of a drop of 10% KOH to vaginal fluid on a slide; 3) vaginal pH greater than 4.5; 4) more than 20% of epithelial cells being clue cells on a vaginal smear slide. Nugent scoring is based on a Gram stain of vaginal fluid smear, with scores of 1-3 being healthy, 4-6 being intermediate; and 7-10 being positive for BV (unhealthy). Note that not all sites may perform Amsel and/or Nugent scoring.

SECONDARY OUTCOMES:
Vaginal pH changes | Baseline, 12 weeks, and 24 weeks will be compared using repeated measures two-way ANOVA with study arm and time as factors.
  The pH of vaginal fluid will be tested using pH test strips. Changes in pH will be compared across time between groups
Vaginal microbiome whole-genome sequencing changes | Baseline to 24 weeks
  The vaginal microbiome will be assessed by whole-genome sequencing. Presence and relative abundance (%) of species/taxa will be reported and used to assign the participant's biome to a Community State Type which will be categorized as healthy, intermediate, or unhealthy (BV). Kruskal-Wallis tests will be used to compare changes in category over time
Vaginal microbiome whole-genome sequencing changes | Baseline to 12 weeks
  The vaginal microbiome will be assessed by whole-genome sequencing. Presence and relative abundance (%) of species/taxa will be reported and used to assign the participant's biome to a Community State Type which will be categorized as healthy, intermediate, or unhealthy (BV). Kruskal-Wallis tests will be used to compare changes in category over time
Vulvovaginal symptoms by questionnaires | Baseline to 24 weeks
  Frequency and intensity of vulvovaginal symptoms will be assessed by questionnaires. The Vulvovaginal Symptoms Questionnaire contains yes/no questions. A proprietary addendum questionnaire uses Likert scale questions where 0 is no symptoms and 3 is severe or very frequent symptoms. Changes over time will be compared between groups using Chi-square for Vulvovaginal Symptoms Questionnaire and Kruskal-Wallis for addendum questions.
Vulvovaginal symptoms by questionnaires | Baseline to 12 weeks
  Frequency and intensity of vulvovaginal symptoms will be assessed by questionnaires. The Vulvovaginal Symptoms Questionnaire contains yes/no questions. A proprietary addendum questionnaire uses Likert scale questions where 0 is no symptoms and 3 is severe or very frequent symptoms. Changes over time will be compared between groups using Chi-square for Vulvovaginal Symptoms Questionnaire and Kruskal-Wallis for addendum questions.

CONTACTS AND LOCATIONS:
Overall Officials: Corey Babb, DO, Principal Investigator — Haven Center for Sexual Medicine & Vulvovaginal Disorders
Locations (1):
- Haven Center for Sexual Medicine & Vulvovaginal Disorders, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Chidawanyika T, Yi CHC, Kelly-Martin R, Cleland J, DuPriest E. Clinical trial to survey results of Flourish vaginal care system for recurrent BV [A80]. Obstet Gynecol. 2022;139:24S. doi:10.1097/01.AOG.0000826648.49549.01
- [Background] O'Hanlon DE, Gajer P, Brotman RM, Ravel J. Asymptomatic Bacterial Vaginosis Is Associated With Depletion of Mature Superficial Cells Shed From the Vaginal Epithelium. Front Cell Infect Microbiol. 2020 Mar 10;10:106. doi: 10.3389/fcimb.2020.00106. eCollection 2020. PMID 32211347
- [Background] Nagot N, Ouedraogo A, Defer MC, Vallo R, Mayaud P, Van de Perre P. Association between bacterial vaginosis and Herpes simplex virus type-2 infection: implications for HIV acquisition studies. Sex Transm Infect. 2007 Aug;83(5):365-8. doi: 10.1136/sti.2007.024794. Epub 2007 May 10. PMID 17493979
- [Background] Denney JM, Culhane JF. Bacterial vaginosis: a problematic infection from both a perinatal and neonatal perspective. Semin Fetal Neonatal Med. 2009 Aug;14(4):200-3. doi: 10.1016/j.siny.2009.01.008. Epub 2009 Apr 11. PMID 19362525
- [Background] Bradshaw CS, Morton AN, Hocking J, Garland SM, Morris MB, Moss LM, Horvath LB, Kuzevska I, Fairley CK. High recurrence rates of bacterial vaginosis over the course of 12 months after oral metronidazole therapy and factors associated with recurrence. J Infect Dis. 2006 Jun 1;193(11):1478-86. doi: 10.1086/503780. Epub 2006 Apr 26. PMID 16652274
- [Background] Sobel JD, Schmitt C, Meriwether C. Long-term follow-up of patients with bacterial vaginosis treated with oral metronidazole and topical clindamycin. J Infect Dis. 1993 Mar;167(3):783-4. doi: 10.1093/infdis/167.3.783. No abstract available. PMID 8440952
- [Background] De Seta F, Campisciano G, Zanotta N, Ricci G, Comar M. The Vaginal Community State Types Microbiome-Immune Network as Key Factor for Bacterial Vaginosis and Aerobic Vaginitis. Front Microbiol. 2019 Oct 30;10:2451. doi: 10.3389/fmicb.2019.02451. eCollection 2019. PMID 31736898
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] Wang Z, He Y, Zheng Y. Probiotics for the Treatment of Bacterial Vaginosis: A Meta-Analysis. Int J Environ Res Public Health. 2019 Oct 12;16(20):3859. doi: 10.3390/ijerph16203859. PMID 31614736
- [Background] Senok AC, Verstraelen H, Temmerman M, Botta GA. Probiotics for the treatment of bacterial vaginosis. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD006289. doi: 10.1002/14651858.CD006289.pub2. PMID 19821358
- [Background] Hallen A, Jarstrand C, Pahlson C. Treatment of bacterial vaginosis with lactobacilli. Sex Transm Dis. 1992 May-Jun;19(3):146-8. doi: 10.1097/00007435-199205000-00007. PMID 1523530
- [Background] Reid G, Burton J, Hammond JA, Bruce AW. Nucleic acid-based diagnosis of bacterial vaginosis and improved management using probiotic lactobacilli. J Med Food. 2004 Summer;7(2):223-8. doi: 10.1089/1096620041224166. PMID 15298771
- [Background] Witkin SS, Mendes-Soares H, Linhares IM, Jayaram A, Ledger WJ, Forney LJ. Influence of vaginal bacteria and D- and L-lactic acid isomers on vaginal extracellular matrix metalloproteinase inducer: implications for protection against upper genital tract infections. mBio. 2013 Aug 6;4(4):e00460-13. doi: 10.1128/mBio.00460-13. PMID 23919998
- [Background] Ananthapadmanabhan KP, Moore DJ, Subramanyan K, Misra M, Meyer F. Cleansing without compromise: the impact of cleansers on the skin barrier and the technology of mild cleansing. Dermatol Ther. 2004;17 Suppl 1:16-25. doi: 10.1111/j.1396-0296.2004.04s1002.x. PMID 14728695
- [Background] France MT, Ma B, Gajer P, Brown S, Humphrys MS, Holm JB, Waetjen LE, Brotman RM, Ravel J. VALENCIA: a nearest centroid classification method for vaginal microbial communities based on composition. Microbiome. 2020 Nov 23;8(1):166. doi: 10.1186/s40168-020-00934-6. PMID 33228810